CLINICAL TRIAL: NCT06033300
Title: Characterization and Quantification of Platelet/Leukocyte Aggregates in Patients With Suspected Heparin-induced Thrombocytopenia
Acronym: HITSTREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2023_843_0047
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Heparin-induced Thrombocytopenia; HIT; Platelet Activation; Platelets; Leukocytes; Platelet/Leukocyte Aggregates; HITSTREAM; Flow Cytometry
Keywords: Heparin-induced Thrombocytopenia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- suspected heparin-induced thrombocytopenia: (Experimental)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — blood sample

SUMMARY:
The investigators would like to analyze platelet/leukoplak activation, quantify and morphologically characterize these aggregates using in vitro analysis, directly on whole blood from adult patients with suspected HIT. This would enable to better describe the in vivo pathophysiology of the HIT-suspect patient, and eliminate the need for platelet donors to perform the usual confirmatory techniques, whose inter- and intra-individual variability is very high. What's more, the SRA test, evaluated as the reference test, requires the use of radioisotopes and is therefore only carried out in a few biological expertise centers, resulting in a very long delay in the delivery of results. It should also be noted that, in practice, HÉPARINE is immediately stopped in patients with suspected HIT, and they are put on an expensive anticoagulant (DANAPAROIDE SODIQUE or ARGATROBAN) in curative doses until the results of the confirmatory tests are back. In this serious, life-threatening condition, it is essential to have a sensitive, specific test to confirm HIT as quickly as possible. Each patient with suspected HIT (rapid >30% reduction in platelet count after initiation of heparin therapy) should have 4 tubes of 3.2% citrated whole blood (2.7ml) collected at the time of suspected HIT (D0) and before any therapeutic switch (or 24 h max after switch). A new sample (4 citrated tubes) will be taken at D4, D7 and D14 during hospitalization, in patients who test positive for anti-PF4/H Ac. All patients with suspected HIT will follow the standard diagnostic pathway, i.e. a screening test (immunological test for anti-PF4/heparin antibodies, total Ig, ACL TOP, Werfen) followed by a confirmatory test (platelet aggregation on TA-8V, STAGO and/or SRA). Doppler ultrasonography of the lower limbs will be performed in HIT-suspect patients with a positive anti-PF4/H antibody test, as currently performed as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Any adult patient suspected of having HIT, with a positive anti-PF4/H antibody test
* Patient signed consent to study participation
* Patient with social security coverage

Exclusion Criteria:

* All adult patients with suspected HIT and negative anti-PF4/H antibody test.
* Protected adults (guardianship, under curators) or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
percentage of CD41a+/CD45- platelet clusters | day 1
  percentage of CD41a+/CD45- platelet clusters relative to platelet count by Flow Imaging ImageStream

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No